CLINICAL TRIAL: NCT06594185
Title: A Prospective, Multicenter, Open Label, Single Arm, Post-Marketing Clinical Study to Evaluate Real World Outcomes of the enVista® Aspire (EA) and Aspire Toric (ETA) Intraocular Lens in Subjects Undergoing Cataract Extraction
Brief Title: A Study to Evaluate Real World Outcomes of the enVista® Aspire (EA) and Aspire Toric (ETA) Intraocular Lens in Subjects Undergoing Cataract Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-SU01-ASRWE-4401
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects bilaterally implanted with enVista Aspire EA or Aspire Toric ETA IOLs (Experimental)
  Interventions: Device: enVista Aspire EA or Aspire Toric ETA IOLs

INTERVENTIONS:
Device: enVista Aspire EA or Aspire Toric ETA IOLs — enVista Aspire EA or Aspire Toric ETA IOLs

SUMMARY:
A study to evaluate the real-world clinical performance of the enVista Aspire and Aspire Toric intraocular lens (IOL) models EA and ETA and to assess surgeon and subject satisfaction

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age or older on the date the Informed Consent Form (ICF) is signed.
2. Subjects must be capable of understanding and providing informed consent on the Institutional Review Board (IRB)- approved Informed Consent Form (ICF) and authorization as appropriate for local privacy regulations.
3. Have a BCDVA at or worse than 20/40 in each eye, with or without a glare source, due to a clinically significant cataract (cortical, nuclear, subcapsular, or combination) that is considered amenable to treatment with standard phacoemulsification cataract extraction and capsular IOL implantation.
4. Have a BCDVA projected to be better than 20/30 after IOL implantation in each eye as determined by the medical judgment of the Principal Investigator.
5. Subjects must have clear intraocular media other than the cataract in both eyes.
6. Subjects must require an IOL power from +6.0 diopter (D) to +34.0 diopter (D) in both eyes.
7. Subjects with clinically significant preoperative corneal astigmatism must require an IOL toric power between 1.25 diopter (D) to 5.75 diopter (D).
8. Subjects must be willing and able to comply with all treatment and follow-up Clinical Investigation visits and procedures

Exclusion Criteria:

1. Pre-existing ocular conditions (subjects with prior corneal refractive surgery, irregular corneal astigmatism, severe (clinically significant) corneal dystrophy, e.g., Fuch's, macular disease, optic nerve atrophy, corneal endothelial disease, abnormal cornea, macular degeneration, retinal degeneration, and chronic drug miosis, who may not achieve the visual acuity of patients without such problems, etc.)
2. Associated ocular conditions that could affect the stability of the IOL (e.g., traumaticzonulolysis, zonular dialysis, evident zonular weakness or dehiscence, etc.) in the study eye.
3. Retinal conditions, or predisposition to retinal conditions, previous history of, or a predisposition to, retinal detachment or proliferative diabetic retinopathy, in which future treatment may be compromised by implanting this IOL
4. Amblyopia
5. Rubella, congenital, traumatic, or complicated cataracts
6. Extremely shallow anterior chamber, not due to swollen cataract
7. Recurrent anterior or posterior segment inflammation of unknown etiology, or any disease producing an inflammatory reaction (e.g., iritis or uveitis)
8. Aniridia
9. Iris neovascularization
10. Subjects who have uncontrolled glaucoma in either eye. Uncontrolled glaucoma is defined as intraocular pressure (IOP) greater than 21 mm Hg in spite of maximally tolerated medications (with more than three topical drugs for IOP control).
11. Microphthalmos or macrophthalmos
12. Previous corneal transplant, prior YAG laser iridotomy, YAG vitreolysis, and prior phakic IOL insertions.
13. Pre-existing ocular conditions that may negatively impact the stability of the implant or intraoperative conditions (posterior capsular rupture, complications in which the IOL stability could be compromised, inability to place IOL in capsular bag, etc.).
14. Mechanical or surgical manipulation required to enlarge the pupil
15. Vitreous loss (significant)
16. Anterior chamber bleeding (significant)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Mean binocular best-corrected distance visual acuity (BCDVA) at Postoperative Visit 1 | Assessed at Postop visit 1 (Day 14 to 42 days after second eye IOL implantation)
  Mean binocular best-corrected distance visual acuity (BCDVA) at Postoperative Visit 1
Percentage of subjects with binocular BCDVA of 20/40 or better at Postoperative Visit 1 | Assessed at Postop visit 1 (Day 14 to 42 days after second eye IOL implantation)
  Percentage of subjects with binocular BCDVA of 20/40 or better at Postoperative Visit 1

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - Site 118, Birmingham, Alabama
  - Site 154, Bullhead City, Arizona
  - Site 137, Chandler, Arizona
  - Site 136, Mesa, Arizona
  - Site 162, Phoenix, Arizona
  - Site 105, Tucson, Arizona
  - Site 104, Bakersfield, California
  - Site 101, Beverly Hills, California
  - Site 151, Hemet, California
  - Site 111, Huntington Beach, California
  - Site 126, Long Beach, California
  - Site 149, Los Angeles, California
  - Site 155, Murrieta, California
  - Site 109, Newport Beach, California
  - Site 112, Orange, California
  - Site 144, Pasadena, California
  - Site 119, Torrance, California
  - Site 115, Upland, California
  - Site 161, Greenwich, Connecticut
  - Site 130, Milford, Connecticut
  - Site 164, Stamford, Connecticut
  - Site 125, Bradenton, Florida
  - Site 148, Mt. Dora, Florida
  - Site 143, Pompano Beach, Florida
  - Site 127, Tarpon Springs, Florida
  - Site 153, Winter Park, Florida
  - Site134, Gainesville, Georgia
  - Site 165, Roswell, Georgia
  - Site 163, Honolulu, Hawaii
  - Site 160, Honolulu, Hawaii
  - Site 108, Rock Island, Illinois
  - Site 133, Shreveport, Louisiana
  - Site 131, Birmingham, Michigan
  - Site 121, Alexandria, Minnesota
  - Site 142, Alexandria, Minnesota
  - Site 102, Bloomington, Minnesota
  - Site 106, Kansas City, Missouri
  - Site 128, Bozeman, Montana
  - Site 117, South Sioux City, Nebraska
  - Site 114, South Orange, New Jersey
  - Site 159, Albuquerque, New Mexico
  - Site132, Poughkeepsie, New York
  - Site 138, Goldsboro, North Carolina
  - Site 156, Leland, North Carolina
  - Site 107, West Fargo, North Dakota
  - Site 103, Brecksville, Ohio
  - Site 129, Cincinnati, Ohio
  - Site 166, Moore, Oklahoma
  - Site 152, Bend, Oregon
  - Site 135, Medford, Oregon
  - Site 150, Allenwood, Pennsylvania
  - Site 140, Bala-Cynwyd, Pennsylvania
  - Site 157, Kingston, Pennsylvania
  - Site 145, Austin, Texas
  - Site 158, Austin, Texas
  - Site 113, Beaumont, Texas
  - Site 110, Dallas, Texas
  - Site 147, Houston, Texas
  - Site 141, Houston, Texas
  - Site 123, San Antonio, Texas
  - Site 124, San Antonio, Texas
  - Site 122, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No